CLINICAL TRIAL: NCT01631955
Title: A Study of Quality of Life and Changes to Symptom Relief for Acute Uncomplicated Cystitis Treated With Antibiotics (Ciprobay); Prospective, Open-label, Multicenter, Observational Study
Brief Title: Assessment of UTI Symptoms and Quality of Life According to Antibiotics Treatment in Acute Uncomplicated Cystitis
Status: Completed | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Kwang-Woo Lee, MD, Department of urology, Soonchunhyang University Hospital
Other Study IDs: KAUTII&Schbc-UTI-QoL
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Acute Cystitis
Keywords: Acute cystitis; Antibiotics; Quality of life

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cystitis: female with cystitis symptoms
  Interventions: Drug: Ciprobay

INTERVENTIONS:
Drug: Ciprobay — Ciprobay (250mg, bid, oral)

SUMMARY:
Although Cystitis includes a clinical syndrome characterized by various combinations of dysuria (painful urination), frequency, urgency, gross haematuria, lower back and/or abdominal/suprapubic discomfort with pyuria and bacteriuria. An acute uncomplicated UTI (referred to as cystitis) has been focused microorganisms and drug-resistance. There has been little research on Clinical aspects on cystitis treatment such as bothersomeness, or the impact of symptoms on patients' quality of life (QoL). The investigators want to study for Assessment of UTI Symptoms and Quality of Life According to Antibiotics Treatment(Ciprobay) in Acute Uncomplicated Cystitis in Korean Women.

ELIGIBILITY:
Inclusion Criteria:

* Female outpatients (20-65 years old)
* Acute cystitis symptoms (subject-reported) for < 1 week prior to Visit 1.

Exclusion Criteria:

* Acute cystitis symptoms for ≥ 1 week prior to Visit 1.
* Diabetes mellitus
* Congenital urinary tract abnormality
* Female subjects who are pregnant, nursing, or with a positive urine pregnancy test or who are intending to become pregnant during the study or within 3 months after the completion of the study.
* Hypersensitivity to the active substance (Ciprobay).
* Subjects who have vaginal discharge
* Fever ( ≥ 37.5 ºC)
* Sexually transmitted diseases.
* Documented significant renal disease (sCr > 1.5)
* Subjects who cannot consent to this study.
* Subjects who had received antimicrobial agents in the previous 4 weeks.
* Recurrent urinary tract infection defined as treatment for UTI > 3 times in the last year.
* Use of an indwelling catheter or an intermittent self-catheterization program.
* Neurogenic bladder.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient
Sampling Method: Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2009-10; Primary Completion 2011-02 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Effect on patient satisfaction and quality of life. | at day 5 relative to baseline

SECONDARY OUTCOMES:
Change in UTISA sub-category (dysuria, frequency, urgency, pain, hematuria) | at day 10, 21 and 28 relative to baseline
Change in KHQ | at day 10, 21 and 28 relative to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Min-Eui Kim, MD, PhD, Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Soonchunhyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do, South Korea